CLINICAL TRIAL: NCT02678390
Title: Stimulating the Production of Ketones Through the Combined Use of Aerobic Exercise (AE) and Dietary a Medium Chain Triglycerides (MCT) Supplement
Brief Title: Medium Chain Triglycerides and Aerobic Exercise on Ketone Production in Women With or Without Prediabetes
Acronym: MCT+AE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2015-508
Record Dates: First submitted 2016-02-05; First posted 2016-02-09 (Estimated); Results first posted 2020-04-07 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-03

CONDITIONS: Prediabetic State
MeSH Terms: conditions — Prediabetic State | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy women (Experimental): Arm: Evaluation of MCT, aerobic exercise alone and MCT+ aerobic exercise on glucose/ketone/lipid/insulin metabolism in 4-hour visits with repeated blood sampling.
  Interventions:
  1. A control day with no MCT and no aerobic exercise.
  2. A 5 day consecutive MCT intake of 30 g/day.
  3. 30 minutes of aerobic exercise at 70% to 80% HRR of intensity.
  4. A 5 day consecutive MCT intake of 30 g/day in combination with 30 minutes of aerobic exercise (70% to 80% HRR)/ day for the five days.
  Interventions: Dietary Supplement: MCT; Dietary Supplement: MCT+ aerobic exercise; Dietary Supplement: Aerobic exercise; Dietary Supplement: Control day
- Women with prediabetes (Experimental): Arm: Evaluation of MCT, aerobic exercise alone and MCT+ aerobic exercise on glucose/ketone/lipid/insulin metabolism in 4-hour visits with repeated blood sampling.
  Interventions:
  1. A control day with no MCT and no aerobic exercise.
  2. A 5 day consecutive MCT intake of 30 g/day.
  3. 30 minutes of aerobic exercise at 70% to 80% HRR of intensity.
  4. A 5 day consecutive MCT intake of 30 g/day in combination with 30 minutes of aerobic exercise (70% to 80% HRR)/ day for the five days.
  Interventions: Dietary Supplement: MCT; Dietary Supplement: MCT+ aerobic exercise; Dietary Supplement: Aerobic exercise; Dietary Supplement: Control day

INTERVENTIONS:
Dietary Supplement: MCT — A 5 day consecutive MCT intake of 30 g/day.
Dietary Supplement: MCT+ aerobic exercise — A 5 day consecutive MCT intake of 30 g/day in combinaison with 30 minutes of aerobic exercise (70% to 80% HRR) per day for the five days.
  Other Names: MCT+AE
Dietary Supplement: Aerobic exercise — A single period of 30 minutes of aerobic exercise (70% to 80% HRR).
  Other Names: AE
Dietary Supplement: Control day — No MCT or aerobic exercise
  Other Names: CTL

SUMMARY:
The aim of this study is to compare the effect on ketone production of dietary an MCT supplement combined or not with physical exercise in two groups of women (N=10/group), healthy adults and patients with prediabetes. After an evaluation of the metabolism (a 4-hour visit with multiple blood samples) at the beginning of the study, all the participants are taken for one-week the MCT supplement alone follow by a one-week period of taking the MCT supplement in combination with physical exercise. At the end of each period of time, the 4-hour visit for the evaluation of the metabolism is repeated.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women group: fasting blood glucose < 6.1 mmol/L and HbA1c < 6.0 %.
* Women with prediabetes: fasting blood glucose between 6.1 and 6.9 mmol/L and HbA1c between 6.0 and 6.4 %

Exclusion Criteria:

* Structured physical activity (more than 2 times per week)
* Inability to practice physical exercise
* Diabetes (fasting glucose ≥ 7.0mmol/L or HbA1c ≥ 6.5%)
* Uncontrolled dyslipidemia or hypertension
* Use of medications known to affect the metabolism of lipids and carbohydrates (steroids, beta-blockers, diuretics, insulin sensitizers, etc.)
* Severe infections or inflammations

Min Age: 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-09; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Cunnane, PhD, Principal Investigator — Research Centre on Aging, CIUSSS de l'Estrie-CHUS
Locations (1):
- Research Centre on Aging - CSSS-IUGS - CIUSSS de l'Estrie - CHUS, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Women; Women With Prediabetes: Arm: Evaluation of MCT, aerobic exercise alone and MCT+ aerobic exercise on glucose/ketone/lipid/insulin metabolism in 4-hour visits with repeated blood sampling.
  Interventions:
  1. A control day with no MCT and no aerobic exercise.
  2. A 5 day consecutive MCT intake of 30 g/day.
  3. 30 minutes of aerobic exercise at 70% to 80% HRR of intensity.
  4. A 5 day consecutive MCT intake of 30 g/day in combination with 30 minutes of aerobic exercise (70% to 80% HRR)/ day for the five days.
  MCT: A 5 day consecutive MCT intake of 30 g/day.
  MCT+ aerobic exercise: A 5 day consecutive MCT intake of 30 g/day in combinaison with 30 minutes of aerobic exercise (70% to 80% HRR) per day for the five days.
  Aerobic exercise: A single period of 30 minutes of aerobic exercise (70% to 80% HRR).
  Control day: No MCT or aerobic exercise
Period: Control (5 Days)
Arm/Group | Healthy Women | Women With Prediabetes
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: MCT (5 Days)
Arm/Group | Healthy Women | Women With Prediabetes
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: AE (1 Day)
Arm/Group | Healthy Women | Women With Prediabetes
Started | 10 | 10
Completed | 10 | 9
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: MCT + AE (5 Days)
Arm/Group | Healthy Women | Women With Prediabetes
Started | 10 | 9
Completed | 10 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Women | Women With Prediabetes | Total
Number analyzed (Participants) | 10 | 9 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (4) | 68 (5) | 68 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 19
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 10 | 9 | 19
Body mass index [Mean (Standard Deviation); unit: kg/m2] | 27 (3) | 28 (4) | 27 (4)
Total body fat [Mean (Standard Deviation); unit: % of body fat] | 43 (6) | 40 (4) | 42 (5)
Plasma glucose [Mean (Standard Deviation); unit: mmol/L] | 5.4 (0.1) | 6.1 (0.4) | 5.8 (0.3)
Glycated hemoglobin [Mean (Standard Deviation); unit: % of glycated hemoglobin] | 5.7 (0.2) | 6.1 (0.2) | 5.9 (0.2)
Ketones [Mean (Standard Deviation); unit: µmol/L] | 153 (94) | 116 (71) | 135 (83)
Triglycerides [Mean (Standard Deviation); unit: mmol/L] | 1.5 (0.4) | 1.6 (0.8) | 1.55 (0.6)
Free Fatty acids [Mean (Standard Deviation); unit: mmol/L] | 0.8 (0.3) | 0.7 (0.3) | 0.75 (0.3)
Insulin [Mean (Standard Deviation); unit: pmol/L] | 64 (11) | 65 (32) | 64.5 (22)

OUTCOME MEASURES:

1. Primary Outcome: Plasma Ketone Concentrations
Description: Acetoacetate (umol/L) and beta-hydroxybutyrate (umol/L); Called Ketones (µmol/L) when combine together The area under the curve (AUC) was calculated according to the trapezoidal method from 0 to 4 h during the visits (interventions) CTL = Metabolic study day (Day 1) MCT = Metabolic study day after 5 days of supplementation (Day 5) AE= Metabolic Study day after acute aerobic exercise (Day 6) AE + MCT = Metabolic Study day after 5 days of aerobic exercise and mct supplementation (Day 11)
Time Frame: 5 days
Measure: Mean (Standard Deviation); unit: (µmol/h)/L
Arm/Group | Healthy Women | Women With Prediabetes
Number analyzed (Participants) | 10 | 9
(µmol/h)/L
  CTL: AUC ketone | -52 (117) | 12 (96)
  MCT: AUC ketone | 493 (243) | 627 (489)
  AE: AUC ketone | 122 (146) | 23 (74)
  MCT+AE: AUC ketone | 835 (444) | 663 (417)

2. Secondary Outcome: Plasma Glucose Concentrations
Description: Glucose (mmol/L) measured in the plasma The area under the curve (AUC) was calculated according to the trapezoidal method from 0 to 4 h during the visits (interventions) CTL = Metabolic study day (Day 1) MCT = Metabolic study day after 5 days of supplementation (Day 5) AE= Metabolic Study day after acute aerobic exercise (Day 6) AE + MCT = Metabolic Study day after 5 days of aerobic exercise and mct supplementation (Day 11)
Time Frame: 5 days
Measure: Mean (Standard Deviation); unit: (mmol*h)/L
Arm/Group | Healthy Women | Women With Prediabetes
Number analyzed (Participants) | 10 | 9
(mmol*h)/L
  CTL: AUC glucose | 7.6 (1.4) | 11.0 (2.8)
  MCT: AUC glucose | 7.3 (1.3) | 11.6 (2.8)
  AE: AUC glucose | 7.6 (1.0) | 10.4 (3.0)
  MCT+AE: AUC glucose | 7.7 (1.5) | 10.3 (1.8)

3. Secondary Outcome: Plasma Triglyceride Concentrations
Description: Triglycerides (mmol/L) measured in the plasma The area under the curve (AUC) was calculated according to the trapezoidal method from 0 to 4 h during the visits (interventions) CTL = Metabolic study day (Day 1) MCT = Metabolic study day after 5 days of supplementation (Day 5) AE= Metabolic Study day after acute aerobic exercise (Day 6) AE + MCT = Metabolic Study day after 5 days of aerobic exercise and mct supplementation (Day 11)
Time Frame: 5 days
Measure: Mean (Standard Deviation); unit: (mmol*h)/L
Arm/Group | Healthy Women | Women With Prediabetes
Number analyzed (Participants) | 10 | 9
(mmol*h)/L
  CTL: AUC triglycerides | 3.6 (0.6) | 3.8 (0.3)
  MCT: AUC triglycerides | 3.9 (0.4) | 3.5 (0.5)
  AE: AUC triglycerides | 4.0 (0.4) | 3.7 (0.7)
  MCT+AE: AUC triglycerides | 3.9 (0.6) | 3.5 (0.8)

4. Secondary Outcome: Plasma Free Fatty Acid Concentrations
Description: Free fatty acids (mmol/L) measured in the plasma The area under the curve (AUC) was calculated according to the trapezoidal method from 0 to 4 h during the visits (interventions) CTL = Metabolic study day (Day 1) MCT = Metabolic study day after 5 days of supplementation (Day 5) AE= Metabolic Study day after acute aerobic exercise (Day 6) AE + MCT = Metabolic Study day after 5 days of aerobic exercise and mct supplementation (Day 11)
Time Frame: 5 days
Measure: Mean (Standard Deviation); unit: (mmol*h)/L
Arm/Group | Healthy Women | Women With Prediabetes
Number analyzed (Participants) | 10 | 9
(mmol*h)/L
  CTL: AUC Free fatty acids | 1.3 (0.3) | 1.3 (0.6)
  MCT: AUC Free fatty acids | 1.3 (0.2) | 1.5 (0.4)
  AE: AUC Free fatty acids | 1.3 (0.2) | 1.4 (0.3)
  MCT+AE: AUC Free fatty acids | 1.4 (0.6) | 1.6 (0.3)

5. Secondary Outcome: Plasma Insulin Concentrations
Description: Insulin (nmol/L) measured in the plasma The area under the curve (AUC) was calculated according to the trapezoidal method from 0 to 4 h during the visits (interventions) CTL = Metabolic study day (Day 1) MCT = Metabolic study day after 5 days of supplementation (Day 5) AE= Metabolic Study day after acute aerobic exercise (Day 6) AE + MCT = Metabolic Study day after 5 days of aerobic exercise and mct supplementation (Day 11)
Time Frame: 5 days
Measure: Mean (Standard Deviation); unit: (nmol*h)/L
Arm/Group | Healthy Women | Women With Prediabetes
Number analyzed (Participants) | 10 | 9
(nmol*h)/L
  CTL: AUC Insulin | 0.9 (0.5) | 0.8 (0.3)
  MCT: AUC Insulin | 0.8 (0.3) | 0.8 (0.8)
  AE: AUC Insulin | 0.8 (0.2) | 0.7 (0.3)
  MCT+AE: AUC Insulin | 0.7 (0.3) | 0.6 (0.2)

ADVERSE EVENTS:
Time Frame: 2 weeks
Arm/Group | Healthy Women | Women With Prediabetes
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/9
Other Adverse Events (participants affected / at risk) | 0/10 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-01): https://cdn.clinicaltrials.gov/large-docs/90/NCT02678390/Prot_SAP_000.pdf